CLINICAL TRIAL: NCT01111851
Title: MK0869 and MK0517 Time-on-Target PET Study
Brief Title: Aprepitant and Fosaprepitant Time-on-Target PET (Positron Emission Tomography) Study (0869-183)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0869-183; 2010_531
Record Dates: First submitted 2010-04-26; First posted 2010-04-28 (Estimated); Results first posted 2011-11-03 (Estimated); Last update posted 2015-02-25 (Estimated); Status verified 2015-02

CONDITIONS: Chemotherapy-Induced Nausea and Vomiting (CINV)
Keywords: NK1-receptor occupancy
MeSH Terms: conditions — Vomiting | interventions — fosaprepitant; Aprepitant; Dexamethasone; Ondansetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fosaprepitant 150 mg (Experimental): Fosaprepitant 150 mg
  Interventions: Drug: Fosaprepitant 150 mg; Drug: Dexamethasone (12-8-16-16 mg); Drug: Ondansetron; Drug: MK0999
- Aprepitant 165 mg (Experimental): Aprepitant 165 mg
  Interventions: Drug: Aprepitant 165 mg; Drug: Dexamethasone (12-8-16-16 mg); Drug: Ondansetron; Drug: MK0999
- Aprepitant 250 mg (Experimental): Aprepitant 250 mg
  Interventions: Drug: Aprepitant 250 mg; Drug: Dexamethasone (12-8-8-16 mg); Drug: Ondansetron; Drug: MK0999

INTERVENTIONS:
Drug: Fosaprepitant 150 mg — a single intravenous infusion of 150 mg fosaprepitant dimeglumine over 20 minutes on Day 1 15 minutes after consumption of a standard light breakfast meal
  Other Names: MK0517
  Arms: Fosaprepitant 150 mg
Drug: Aprepitant 165 mg — a single oral 165 mg aprepitant capsule 15 minutes after consumption of a standard light breakfast meal
  Other Names: MK0869
  Arms: Aprepitant 165 mg
Drug: Aprepitant 250 mg — a single oral 250 mg dose achieved by administering two 125 mg aprepitant capsules 15 minutes after consumption of a standard light breakfast meal
  Other Names: MK0869
  Arms: Aprepitant 250 mg
Drug: Dexamethasone (12-8-16-16 mg) — Dexamethasone 12 mg will be administered orally 30 minutes after the start of fosaprepitant dimeglumine or 30 minutes after aprepitant on Day 1; Oral doses of dexamethasone will be administered on Day 2 (8 mg), Day 3 (8 mg twice daily), and Day 4 (8 mg twice daily) with or without a meal.
  Other Names: Dexamethasone
  Arms: Aprepitant 165 mg; Fosaprepitant 150 mg
Drug: Dexamethasone (12-8-8-16 mg) — Dexamethasone 12 mg will be administered orally 30 minutes after after aprepitant on Day 1; Oral doses of dexamethasone will be administered on Day 2 (8 mg), Day 3 (8 mg), and Day 4 (8 mg twice daily) with or without a meal.
  Other Names: Dexamethasone
  Arms: Aprepitant 250 mg
Drug: Ondansetron — The intravenous (I.V.) infusion of ondansetron 32 mg will begin 30 minutes after the start of fosaprepitant dimeglumine or 30 minutes after aprepitant on Day 1 and will be administered as a 15-minute infusion
Drug: MK0999 — I.V. infusion of MK0999 containing ~100 MBq (~3 mCi) containing ≤ 5 ug of MK0999)

SUMMARY:
This study will evaluate if the mean value of brain neurokinin 1 (NK1)-receptor occupancy of participants treated with aprepitant is similar to that of participants treated with fosaprepitant at certain timepoints.

DETAILED DESCRIPTION:
The third arm of the study (Aprepitant 250 mg) will only be conducted if the real-time assessment of the NK1-receptor occupancy data between fosaprepitant 150 mg & aprepitant 165 mg reveals that the primary hypothesis will not be supported.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy
* Female participants must be of non-childbearing potential
* Non-smoker or has not used nicotine or nicotine-containing products for at least 6 months

Exclusion Criteria:

* History of a clinically significant psychiatric disorder over the last 5 to 10 years
* History of stroke, chronic seizures, or major neurological disorder
* History of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases
* History of neoplastic disease
* Excessive consumption of alcohol (3 drinks/day) or caffeinated beverages (6 servings/day)
* Major surgery, donated or lost 1 unit of blood within 4 weeks
* Participated in another investigational study within 4 weeks
* History of significant drug allergy or any clinically significant adverse

experiences related to EMEND™, dexamethasone, or ondansetron

* History of significant multiple and/or severe allergies
* History of anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food
* Current drug/alcohol abuse, or history of such within 2 years
* Participation in a PET study or other study involving administration of a radioactive substance or ionizing radiation within the prior 12 months
* Extensive radiological examination within the prior 12 months
* Magnetizable metal prostheses or devices (Magnetic Resonance Imaging (MRI) hazard)
* History of claustrophobia

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2010-04; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Van Laere K, De Hoon J, Bormans G, Koole M, Derdelinckx I, De Lepeleire I, Declercq R, Sanabria Bohorquez SM, Hamill T, Mozley PD, Tatosian D, Xie W, Liu Y, Liu F, Zappacosta P, Mahon C, Butterfield KL, Rosen LB, Murphy MG, Hargreaves RJ, Wagner JA, Shadle CR. Equivalent dynamic human brain NK1-receptor occupancy following single-dose i.v. fosaprepitant vs. oral aprepitant as assessed by PET imaging. Clin Pharmacol Ther. 2012 Aug;92(2):243-50. doi: 10.1038/clpt.2012.62. Epub 2012 Jun 27. PMID 22739139

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Aprepitant 250 mg was not evaluated because the assessment of the positron emission tomography (PET) scan data (neurokinin 1 (NK1)-receptor occupancy values at 24 & 48 hours postdose) from fosaprepitant 150 mg & aprepitant 165 mg revealed that the protocol's hypothesis was met; therefore, it was not necessary to evaluate aprepitant 250 mg.
Groups:
- Fosaprepitant 150 mg: A single intravenous infusion of 150 mg fosaprepitant dimeglumine over 20 minutes, 15 minutes after consumption of a standard light breakfast meal on Day 1.
- Aprepitant 165 mg: A single oral 165 mg aprepitant capsule 15 minutes after consumption of a standard light breakfast meal on Day 1.
Period: Overall Study
Arm/Group | Fosaprepitant 150 mg | Aprepitant 165 mg
Started | 8 | 8
Completed | 6 | 8
Not Completed | 2 | 0
Not completed — All planned PET scans were not obtained. | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fosaprepitant 150 mg | Aprepitant 165 mg | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Customized [Number; unit: Participants]
  < = 18 years | 0 | 0 | 0
  Between 18 and 55 years | 8 | 8 | 16
  > = 55 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 8 | 16
Region of Enrollment [Number; unit: participants]
  Belgium | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Brain NK1-receptor Occupancy at 24 Hours Post Dose
Time Frame: 24 hours post dose
Population: All participants with at least 1 successful post dose PET
  scan were included in the analysis population.
Measure: Geometric Mean (95% Confidence Interval); unit: Percent of occupancy
Arm/Group | Fosaprepitant 150 mg | Aprepitant 165 mg
Number analyzed (Participants) | 5 | 5
Percent of occupancy | 100.40 [99.51 to 101.29] | 100.20 [99.31 to 101.09]
Statistical Analysis 1: Comparison: Fosaprepitant 150 mg vs Aprepitant 165 mg; Test type: Superiority or Other; Geometric Mean Ratio of the LS Means = 1.00, 90% CI 2-sided [0.99 to 1.01] — The point estimate and 90% confidence interval (CI) were generated for the geometric mean ratio (GMR) [aprepitant 165 mg/fosaprepitant 150 mg]

2. Primary Outcome: Brain NK1-receptor Occupancy at 48 Hours Post Dose
Time Frame: 48 hours post dose
Population: All participants with at least 1 successful postdose PET
  scan were included in the analysis population.
Measure: Geometric Mean (95% Confidence Interval); unit: Percent of occupancy
Arm/Group | Fosaprepitant 150 mg | Aprepitant 165 mg
Number analyzed (Participants) | 4 | 5
Percent of occupancy | 98.62 [96.91 to 100.37] | 98.79 [97.19 to 100.42]
Statistical Analysis 1: Comparison: Fosaprepitant 150 mg vs Aprepitant 165 mg; Test type: Superiority or Other; Geometric Mean Ratio of the LS means = 1.00, 90% CI 2-sided [0.98 to 1.02] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Brain NK1-receptor Occupancy at the Time of the Maximum Concentration (Tmax)
Time Frame: 30 minutes after the end of the 20-minute infusion of fosaprepitant or at 4 hours after oral dosing of aprepitant
Population: All participants with at least 1 successful postdose PET
  scan were included in the analysis population.
Measure: Geometric Mean (95% Confidence Interval); unit: Percent of occupancy
Arm/Group | Fosaprepitant 150 mg | Aprepitant 165 mg
Number analyzed (Participants) | 2 | 3
Percent of occupancy | 100.25 [97.22 to 103.39] | 99.99 [97.47 to 102.58]
Statistical Analysis 1: Comparison: Fosaprepitant 150 mg vs Aprepitant 165 mg; Test type: Superiority or Other; Geometric Mean Ratio of the LS means = 1.00, 90% CI 2-sided [0.97 to 1.03] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Brain NK1-receptor Occupancy at 120 Hours Post Dose
Time Frame: 120 hours post dose
Population: All participants with at least 1 successful postdose PET
  scan were included in the analysis population.
Measure: Geometric Mean (95% Confidence Interval); unit: Percent of occupancy
Arm/Group | Fosaprepitant 150 mg | Aprepitant 165 mg
Number analyzed (Participants) | 3 | 3
Percent of occupancy | 59.93 [34.37 to 104.49] | 54.32 [31.15 to 94.71]
Statistical Analysis 1: Comparison: Fosaprepitant 150 mg vs Aprepitant 165 mg; Test type: Superiority or Other; Geometric Mean Ratio of the LS means = 0.91, 90% CI 2-sided [0.50 to 1.66] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Arm/Group | Fosaprepitant 150 mg | Aprepitant 165 mg
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 5/8 | 8/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fosaprepitant 150 mg (N=8) | Aprepitant 165 mg (N=8)
Vision blurred (Eye disorders) | 1 | 1
Visual impairment (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 4
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 4
Fatigue (General disorders) | 0 | 1
Influenza like illness (General disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Positron emission tomogram abnormal (Investigations) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 1
Dizziness postural (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Flushing (Vascular disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication guidelines.